CLINICAL TRIAL: NCT03812458
Title: Impact of the Guidance, Through Website and Brochure, in the Symptoms of Acute Stress and Anxiety in Relatives of Critically Ill Paciente in Intensive Care Unit: Randomized Clinical Trial
Brief Title: GASA-CIR Trail (Guidance and the Symptoms of Acute Stress and Anxiety in Critically Ill Patients Relatives in Intensive Care Unit)
Acronym: GASA-CIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital Moinhos de Vento (Other); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Vitória Homem Machado, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: acute stress,anxiety
Record Dates: First submitted 2018-11-05; First posted 2019-01-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Acute Stress Disorder; Anxiety; Depression
Keywords: resilience; anxiety; acute stress; relatives; critical ill patients
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Parallel multicentric randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidance (Experimental): The intervention group will consist of the relatives who will receive a printed brochure and are encouraged to visit a website with detailed information and with simple language regarding the ICU environment (treatments, care, alarms, multidisciplinary team) and the characteristics of critically ill patients (organ dysfunction, prognosis, palliative care, organ dysfunction).
  Interventions: Behavioral: website and brochure
- Control (No Intervention): The families who will not receive the brochure and are not encouraged to visit the website.

INTERVENTIONS:
Behavioral: website and brochure — website and brochure
  Arms: Guidance

SUMMARY:
A randomized clinical trial 1:1 among relatives of patients admitted to an intensive care unit, the intervention group will be composed by family members who receive a printed brochure and will be encouraged to visit a website detailed information and plain language about the ICU environment and the critically ill patient characteristics. The primary outcome will be the impact of orientations on symptoms of post-traumatic stress, assessed by the IES-R scale. Secondary outcome measures will include symptoms of anxiety and depression at the end of 7 days and after 3 months of follow-up by the HADS scales, the degree of satisfaction of the relatives, through the FS-ICU scale, as well as the association of resilience, through the CD-RISC scale, with the symptoms of anxiety and depression.

DETAILED DESCRIPTION:
The hospitalization of one family member may be responsible for the generation of anxiety and depression, especially if the patient environment for the intensive care unit (ICU). The orientation of family members, through website and brochure, seems to have effect of reducing these symptoms, however, there is a shortage of studies capable of such conduct. The focus of this study will be to evaluate the impact of family guidance in reducing symptoms of depression, acute stress and anxiety displayed by them, in addition to verifying the association between resilience.

A randomized clinical trial 1:1 among relatives of patients admitted to an intensive care unit, the randomization will be in blocks of different sizes and stratified according to the educational level of the familiar. Intervention group will be composed by family members who receive a printed brochure and will be encouraged to visit a website detailed information and plain language about the ICU environment (treatments, care, alarms, multidisciplinary team) and the critically ill patient characteristics (organic dysfunction, prognosis, palliative care, organ dysfunction). The family, of the control group, will not receive the printed brochure and are not encouraged to visit the website. After hospitalization of the patient in the ICU, the research team will have up to 48 hrs to evaluate the eligibility criteria of the next of kin of this patient. Primary outcome will be the impact of orientations on symptoms of post-traumatic stress, assessed by the IES-R scale. Secondary outcome measures will include symptoms of anxiety and depression at the end of 7 days and after 3 months of follow-up by the HADS scale, the degree of satisfaction of the relatives, through the FS-ICU scale, as well as the association of resilience, through the CD-RISC scale, with the symptoms of anxiety and depression The study will occur with families of patients admitted to the ICUs of Hospital Moinhos de Vento and Hospital Ernesto Dornelles. We will collect characteristics related to demographic, social, educational features, levels of resilience, religiosity and prior history of mood disorder, anxiety disorder or post-traumatic stress disorder, length of ICU stay, SAPS III, and ICU and hospital outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For patient, with more than 18 years old, who ICU admission exceeding 48 hours;
* For Patient's Family Members: familiar close to a patient hospitalized in the ICU (spouse, father, mother, son, daughter, grandmother, brother, sister, uncle, aunt, cousin);

Exclusion Criteria:

- For Patient's Family Members: communication difficulty (illiteracy, not speaking Portuguese, deafness or mutism). Some other family member of the patient has already been included in the study. Refusal to sign the term of free and clarified consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Acute stress in critically ill relatives. | After 7 days from enrollment in ICU.
  Using the Impact of Events Scale-Revised. The scale contains 22 questions. It evaluates the subjective distress caused by traumatic events. Items are rated on a 5-point scale, ranging from 0 (nothing) to 4 (extremely). The total score ranges from 0 to 88. A score greater than 33 identifies individuals with symptoms of acute stress disorder.

SECONDARY OUTCOMES:
Satisfaction of the relatives of patients admitted to the ICU: FS-ICU scale | After 7 days from enrollment in ICU.
  Using the FS-ICU scale. The Family Satisfaction in the Intensive Care Unit (FS-ICU) questionnaire measures family satisfaction with care in the intensive care unit. The score ranges 0-100, with higher scores indicating greater satisfaction.
Symptoms of post-traumatic stress. | 3 months from enrollment in ICU.
  Assessed by the Impact of Events Scale-Revised (IES-R). The scale contains 22 questions. It evaluates the subjective distress caused by traumatic events. Items are rated on a 5-point scale, ranging from 0 (nothing) to 4 (extremely). The total score ranges from 0 to 88. A score greater than 33 identifies individuals with symptoms of acute stress disorder.
Symptoms of anxiety and depression | 3 months from enrollment in ICU.
  Using the HADS scale. The questionnaire is composed of 14 questions. The total score ranges from 0 to 42. Score greater than 8 in subgroup, or a total score greater than 16, identify patients with anxiety and depression symptoms.
Symptoms of anxiety and depression | After 7 days from enrollment in ICU.
  Using the HADS scale. The questionnaire is composed of 14 questions. The total score ranges from 0 to 42. Score greater than 8 in subgroup, or a total score greater than 16, identify patients with anxiety and depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No